CLINICAL TRIAL: NCT00638391
Title: Postmenopausal Women With Early Hormone-Receptor Positive Breast Cancer/no Metastasis
Brief Title: Ax-003/Arimidex (Anastrozole) in the Adjuvant Therapy of Early Breast Cancer
Acronym: Ax-003
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar - Medical Science Director, AstraZeneca
Other Study IDs: Ax-003; Ax-003/Arimidex
Record Dates: First submitted 2008-03-13; First posted 2008-03-19 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Breast Cancer
Keywords: Primary early MCa; Arimidex
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all patients treated with Anastrozole
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole
  Other Names: Arimidex

SUMMARY:
The purpose of this study is the initial/followed by 5 year adjuvant therapy with Anastrozole.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with early hormone receptor positive breast cancer/no metastasis

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2005-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
evaluation of Anastrozole therapy as adjuvant treatment in post.menopausal women with not advanced breast cancer únder naturalistic conditions | 12 months

SECONDARY OUTCOMES:
description of population treated with anastrozole | 12 months
further information about the change of specific laboratory parameters | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: H Brasch, Study Director — AstraZeneca Germany